CLINICAL TRIAL: NCT02415036
Title: An International Multi-center Phase 2 Study to Evaluate the Efficacy and Safety of Melphalan Hydrochloride for Injection for Use With the Hepatic Delivery System Treatment in Patients With Unresectable Hepatocellular Carcinoma or Intra Hepatic Cholangiocarcinoma
Brief Title: Melphalan for Use With the Hepatic Delivery System Treatment in Patients With Unresectable Hepatocellular Carcinoma or Intra Hepatic Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited enrollment
Sponsor: Delcath Systems Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHP-HCC-202
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Hepatocellular Carcinoma; Intrahepatic Cholangiocarcinoma
Keywords: HCC; ICC; Percutaneous hepatic perfusion
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma | interventions — Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Melphalan/HDS treatment of patients with HCC (Experimental): Percutaneous hepatic perfusion with melphalan hydrochloride for injection using the Hepatic Delivery System on patients with Hepatocellular carcinoma (HCC).
  Melphalan hydrochloride is administered at a dose of 3mg/kg ideal body weight once every 6 weeks for a maximum of 2 cycles of treatment.
  Interventions: Device: Delcath Hepatic Delivery System; Drug: Melphalan
- Melphalan/HDS treatment of patients with ICC (Experimental): Percutaneous hepatic perfusion with melphalan hydrochloride for injection using the Hepatic Delivery System on patients with Intrahepatic cholangiocarcinoma (ICC).
  Melphalan hydrochloride is administered at a dose of 3mg/kg ideal body weight once every 6 weeks for a maximum of 2 cycles of treatment.
  Interventions: Device: Delcath Hepatic Delivery System; Drug: Melphalan

INTERVENTIONS:
Device: Delcath Hepatic Delivery System
  Other Names: Melphalan/Hepatic Delivery System; Percutaneous hepatic perfusion (PHP)
Drug: Melphalan

SUMMARY:
This is a two arm, open label, multi-center, Phase 2 study to evaluate the efficacy and safety of Melphalan/HDS in patients with unresectable Hepatocellular Carcinoma (HCC) or Intra Hepatic Cholangiocarcinoma (ICC) confined to the liver.

DETAILED DESCRIPTION:
This is a two arm, open label, multi-center, Phase 2 study to evaluate the efficacy and safety of Melphalan/HDS in patients with unresectable HCC or ICC confined to the liver.

Eligible patients will receive up to 2 Melphalan/HDS treatments. Each treatment cycle consists of 6 weeks with an acceptable delay for another 2 weeks before next planned treatment. Tumor response will be assessed at the end of cycle 2.

The Melphalan/HDS treatment will be terminated in patients with progressive disease (PD) after the 1st treatment and based on safety in patients with > 8 weeks delay of recovery from toxicity.

ELIGIBILITY:
Inclusion Criteria:

Patients with HCC must meet all of the following criteria for study entry:

1. HCC diagnosed by tissue or imaging study.
2. Unresectable HCC without clinically significant extra hepatic disease (minor lesions [≤ 1 cm and not consistent with metastatic disease] acceptable) based on computed tomography (CT).
3. At least one target lesion based on mRECIST. In patients with prior loco-regional therapy, the target lesion(s) must be located in area(s) outside previous treatment or must have progressed after prior treatment if located within previous treatment field.
4. Child-Pugh Class A.
5. ECOG PS 0-1.
6. No prior radiation therapy to the liver including Y90-, I131-based loco-regional therapy. Prior loco regional therapy, including resection, based on other technology for HCC, if any, must have been completed at least 4 weeks prior to baseline imaging.
7. Age ≥ 18 years.
8. Signed informed consent.

Patients with ICC must meet all of the following criteria for study entry:

1. ICC diagnosed by tissue or imaging study.
2. Unresectable ICC without clinically significant extra hepatic disease (minor lesions [≤ 1 cm and not consistent with metastatic disease] acceptable) based on CT.
3. At least one target lesion based on mRECIST. In patients with prior loco regional therapy, the target lesion(s) must be located in area(s) outside previous treatment or must have progressed after prior treatment if located within previous treatment field.
4. Child-Pugh Class A.
5. ECOG PS 0-1.
6. No prior radiation therapy to the liver including Y90 , I131 based loco regional therapy. Prior loco regional therapy, including resection, based on other technology for ICC, if any, must have been completed at least 4 weeks prior to baseline imaging.
7. Age ≥ 18 years.
8. Signed informed consent.

Exclusion Criteria:

For the HCC cohort, patients for whom transplantation, radiofrequency ablation (RFA), transarterial chemoembolization (TACE), or systemic treatment with sorafenib are better therapeutic options are to be excluded from study entry.

Additionally, for both the HCC and ICC cohorts, patients who meet any of the following criteria will be excluded from study entry:

1. Greater than 50% tumor burden in the liver by imaging.
2. History of orthotopic liver transplantation, Whipple's procedure, hepatic vasculature incompatible with perfusion, hepatofugal flow in the portal vein or known unresolved venous shunting.
3. Evidence of ascites on imaging study, or the use of diuretics for ascites.
4. Clinically significant encephalopathy.
5. History of, or known, hypersensitivity to any components of melphalan or the components of the Melphalan/HDS system.
6. Known hypersensitivity to heparin or the presence of heparin-induced thrombocytopenia.
7. Received an investigational agent for any indication within 30 days prior to first treatment.
8. Not recovered from side effects of prior therapy to ≤ Grade 1 (according to National Cancer Institute [NCI] CTCAE version 4.03). Certain side effects that are unlikely to develop into serious or life-threatening events (e.g. alopecia) are allowed at > Grade 1.
9. Those with New York Heart Association functional classification II, III or IV; active cardiac conditions including unstable coronary syndromes (unstable or severe angina, recent myocardial infarction), worsening or new-onset congestive heart failure, significant arrhythmias and severe valvular disease must be evaluated for risks of undergoing general anesthesia.
10. History or evidence of clinically significant pulmonary disease that precludes the use of general anesthesia.
11. Uncontrolled diabetes mellitus, hypothyroidism, or hyperthyroidism.
12. Active infection, including Hepatitis B and Hepatitis C infection. Patients with anti-hepatitis B core antigen (HBc) positive, or hepatitis B surface antigen (HBsAg) but viral deoxyribonucleic acid (DNA) negative are exception(s).
13. History of bleeding disorders.
14. Brain lesions with a propensity to bleed.
15. Known varices at risk of bleeding, including medium or large esophageal or gastric varices, or active peptic ulcer.
16. Previous malignancy within 3 years prior to enrollment, except for curatively-treated basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, bladder carcinoma in situ or breast cancer in situ.
17. Inadequate hematologic function as evidenced by any of the following:

    1. Platelets < 90,000/µL
    2. Hemoglobin < 8 g/dL, independent of transfusion or growth factor support
    3. Neutrophils < 1,500 cells/µL.
18. Serum creatinine > 1.5 mg/dL.
19. Inadequate liver function as evidenced by any of the following:

    1. Total serum bilirubin ≥ 2.0 mg/dL
    2. Prothrombin time (PT)/international normalized ratio (INR) > 1.5
    3. Aspartate aminotransferase (AST) > 10 times the upper limit of normal (ULN) or alanine aminotransferase (ALT) > 5 times ULN
    4. Serum albumin < 3.0 g/dL.
20. Known alcohol abuse.
21. For female subjects of childbearing potential (i.e., have had a menstrual period within the past 12 months): a positive serum pregnancy test (β-human chorionic gonadotropin [β HCG]) within 7 days prior to enrollment; or unwilling or unable to undergo hormonal suppression to avoid menstruation during treatment.
22. Sexually active females of childbearing potential and sexually active males with partners of reproductive potential: unwilling or unable to use appropriate contraception from screening until at least 30 days after last administration of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-06; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Objective response rate in percentage of Melphalan/HDS treatment | 2 years

SECONDARY OUTCOMES:
Number of patients with adverse events after treatment with Melphalan/HDS. | 2 years
Progression free survival in months of patients receiving Melphalan/HDS treatment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Johnny John, MD, Study Director — Delcath Systems
Locations (3):
- Germany (3):
  - Universitätsklinikum Frankfurt, Frankfurt
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena